CLINICAL TRIAL: NCT00023933
Title: Phase I Trial of 131I-HuCC49^CH2 for Colon Cancer
Brief Title: Radiolabeled Monoclonal Antibody Therapy in Treating Patients With Recurrent or Persistent Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02406; UAB 9846; CDR0000068877 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-09-13; First posted 2003-06-20 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Adenocarcinoma of the Colon; Adenocarcinoma of the Rectum; Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

ARMS (1):
- Treatment (monoclonal antibody) (Experimental): Patients receive a tracer dose of iodine I 131 monoclonal antibody CC49-deltaCH2 IV on day 1 and a therapy dose over 30 minutes on day 8.
  Cohorts of 3-5 patients receive escalating doses of iodine I 131 monoclonal antibody CC49-deltaCH2 until the MTD is determined. The MTD is defined as the dose at which 3 of 5 patients experience grade 3 or greater toxicity while 0-2 of 5 patients experience reversible grade 4 hematologic toxicity.
  Interventions: Drug: iodine I 131 monoclonal antibody CC49-deltaCH2

INTERVENTIONS:
Drug: iodine I 131 monoclonal antibody CC49-deltaCH2 — Given IV
  Other Names: 131I-HuCC49-deltaCH2; 131I-MOAB CC49-deltaCH2

SUMMARY:
Phase I trial to study the effectiveness of radiolabeled monoclonal antibody therapy in treating patients who have recurrent or persistent metastatic colorectal cancer. Radiolabeled monoclonal antibodies can locate tumor cells and deliver tumor-killing substances to them without harming normal cells. Radiolabeled monoclonal antibody therapy may be effective treatment for colorectal cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of iodine I 131 monoclonal antibody CC49-deltaCH2 (deleted CH2 region) in patients with colorectal cancer.

II. Determine the toxic effects, plasma pharmacokinetics, whole body biodistribution, and conjugate stability of this drug in these patients.

III. Determine the ability of this drug to localize to tumor sites in these patients.

IV. Determine the immune response in patients treated with this drug.

OUTLINE: This is a dose-escalation study.

Patients receive a tracer dose of iodine I 131 monoclonal antibody CC49-deltaCH2 IV on day 1 and a therapy dose over 30 minutes on day 8.

Cohorts of 3-5 patients receive escalating doses of iodine I 131 monoclonal antibody CC49-deltaCH2 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 3 of 5 patients experience grade 3 or greater toxicity while 0-2 of 5 patients experience reversible grade 4 hematologic toxicity.

Patients are followed weekly for a minimum of 7 weeks and then every 6 weeks until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic adenocarcinoma of the colon or rectum

  * Not amenable to surgical resection
  * Recurrent or persistent disease after standard surgery, radiotherapy, and chemotherapy, including fluorouracil and irinotecan
* TAG-72 positive
* Performance status - ECOG 0-2
* WBC greater than 3,500/mm^3
* Platelet count greater than 125,000/mm^3
* Hemoglobin greater than 10 g/dL
* No nucleated RBC or significant teardrop RBC morphology
* Bilirubin less than 1.5 mg/dL
* SGOT/SGPT less than 4 times normal
* Hepatitis B surface antigen negative
* Creatinine less than 2.0 mg/dL
* HIV negative
* No other malignancy within the past 5 years except basal cell skin cancer
* No allergy to iodine
* No detectable antibody to monoclonal antibody CC49
* Not pregnant or nursing
* Fertile patients must use effective contraception
* At least 3 weeks since prior immunotherapy and recovered
* No prior bone marrow or stem cell transplantation
* No other concurrent immunotherapy
* See Disease Characteristics
* At least 3 weeks since prior chemotherapy and recovered
* No concurrent chemotherapy
* See Disease Characteristics
* At least 3 weeks since prior radiotherapy and recovered
* No prior radiotherapy to more than 25% of red marrow
* No concurrent radiotherapy
* See Disease Characteristics
* At least 3 weeks since prior surgery and recovered

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2001-10; Primary Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of 131I-HuCC49^CH2 based on dose-limiting toxicities | 6 weeks

SECONDARY OUTCOMES:
Immune response | Up to 54 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ruby Meredith, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States